CLINICAL TRIAL: NCT04561999
Title: Value of Ultrasound Elastography in Characterization of Superficial Lymphadenopathy
Brief Title: Elastography in Superficial Lymphadenopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermin Gamal Eldin Ahmed Abdel Sattar, Principal investigator, Assiut University
Other Study IDs: Ultrasound in Lymphadenopathy
Record Dates: First submitted 2020-09-14; First posted 2020-09-24 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Superficial Lymphadenopathy
MeSH Terms: interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Superficial Lymphadenopathy
  Interventions: Device: Elastography

INTERVENTIONS:
Device: Elastography — Performance of Ultrasound, Elastography

SUMMARY:
Evaluation of the role of Ultrasound Elastography in differentiation between benign and malignant lymph nodes and its additional information over the classic gray scale and color Doppler ultrasound.

DETAILED DESCRIPTION:
Lymph nodes are part of the body immune system which are located throughout the body including head and neck, armpit, and groin.

Lymphadenopathy is defined as an abnormality in the size or character of lymph nodes caused by the invasion or propagation of either inflammatory or neoplastic cells into the nodes.

The differentiation of malignant from benign lymph nodes is essential because it predicts the patient prognosis and help in the decision making regarding the management plan.

On ultrasound, gray scale sonography helps to evaluate nodal morphology, whilst color doppler is used to assess vascular pattern. The qualitative criteria for malignancy were heterogenous hypoechoic cortex, irregular margins, lack of hyperechoic fatty hilum and abnormal blood vessels penetrating the lymph nodes capsule.The avascular or hilar patterns were defined as LNs with normal vascularity pattern, and the peripheral or mixed (peripheral and hilar) pattern as LNs with abnormal vascularity pattern. On B-mode and color doppler ultrasound, there is no specific criteria for differentiating metastatic lymph nodes from reactive lymph nodes with 100% accuracy.

Fine-needle aspiration biopsy is the reference standard for differentiating metastatic lymph nodes from reactive lymph nodes. However, restrictions of fine-needle aspiration biopsy are that it is an invasive procedure, and it is not possible to perform for lymph nodes smaller than 5 mm.Therefore, a simple, reliable, and non-invasive imaging modality for differentiating malignant lymph nodes is required.

Ultrasound elastography (UE) is a rather new, non-invasive imaging technique that can be used to depict tissue stiffness and elastic properties. Ultrasound elastography (UE) can be divided broadly into 2 groups depending on the type of tissue displacement:

1. Strain elastography (SE): measures tissue displacements along the axis of an applied force.Strain elastography provides semi - quantitative scores based on elastographic pattern (scores based on percentage of stiff area within the lesion) and strain ratio (ratio between the lesion and the background tissue).
2. Shear wave elastography (SWE): measures a different type of waves that is also produced when tissues are mechanically stimulated. Shear wave elastography is also a quantitative method of analysis for elasticity images using shear wave speed (m/s) or elastic modulus (kPa).

Ultrasound elastography (UE) is easy, rather cheap, non-invasive, and quick to perform, well tolerated by patients, and offers a strong diagnostic power.

ELIGIBILITY:
Inclusion Criteria:

• Patients presented with enlarged lymph nodes by clinical examination.

Exclusion Criteria:

* Patients who previously receive any medical treatment or chemo or radiotherapy.
* Patients who previously underwent fine needle aspiration cytology or biopsy.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with enlarged lymph nodes.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the role of Ultrasound Elastography in differentiation between benign and malignant lymph nodes by its additional information over the classic gray scale and color Doppler ultrasound. | one year
  Strain elastography (SE): measures tissue displacements along the axis of an applied force. Strain elastography provides semi - quantitative scores based on elastographic pattern (scores based on percentage of stiff area within the lesion) and strain ratio (ratio between the lesion and the background tissue).
To evaluate the role of Ultrasound Elastography in differentiation between benign and malignant lymph nodes by its additional information over the classic gray scale and color Doppler ultrasound. | one year
  Shear wave elastography (SWE): measures a different type of waves that is also produced when tissues are mechanically stimulated. Shear wave elastography is also a quantitative method of analysis for elasticity images using shear wave speed (m/s).

REFERENCES:
- [Background] Kilic A, Colakoglu Er H. Virtual touch tissue imaging quantification shear wave elastography for determining benign versus malignant cervical lymph nodes: a comparison with conventional ultrasound. Diagn Interv Radiol. 2019 Mar;25(2):114-121. doi: 10.5152/dir.2019.18406. PMID 30774094
- [Background] Acu L, Oktar SO, Acu R, Yucel C, Cebeci S. Value of Ultrasound Elastography in the Differential Diagnosis of Cervical Lymph Nodes: A Comparative Study With B-mode and Color Doppler Sonography. J Ultrasound Med. 2016 Nov;35(11):2491-2499. doi: 10.7863/ultra.15.09019. PMID 27794132
- [Background] Naik RM, Pai A, Guruprasad Y, Singh R. Efficacy of colour Doppler ultrasound in diagnosis of cervical lymphadenopathy. J Maxillofac Oral Surg. 2013 Jun;12(2):123-9. doi: 10.1007/s12663-012-0395-1. Epub 2012 Aug 24. PMID 24431828
- [Background] Suh CH, Choi YJ, Baek JH, Lee JH. The diagnostic performance of shear wave elastography for malignant cervical lymph nodes: A systematic review and meta-analysis. Eur Radiol. 2017 Jan;27(1):222-230. doi: 10.1007/s00330-016-4378-3. Epub 2016 May 5. PMID 27147221
- [Background] Desmots F, Fakhry N, Mancini J, Reyre A, Vidal V, Jacquier A, Santini L, Moulin G, Varoquaux A. Shear Wave Elastography in Head and Neck Lymph Node Assessment: Image Quality and Diagnostic Impact Compared with B-Mode and Doppler Ultrasonography. Ultrasound Med Biol. 2016 Feb;42(2):387-98. doi: 10.1016/j.ultrasmedbio.2015.10.019. Epub 2015 Nov 23. PMID 26617244
- [Background] Bhatia KS, Lee YY, Yuen EH, Ahuja AT. Ultrasound elastography in the head and neck. Part I. Basic principles and practical aspects. Cancer Imaging. 2013 Jul 22;13(2):253-9. doi: 10.1102/1470-7330.2013.0026. PMID 23876352
- [Background] Cheng KL, Choi YJ, Shim WH, Lee JH, Baek JH. Virtual Touch Tissue Imaging Quantification Shear Wave Elastography: Prospective Assessment of Cervical Lymph Nodes. Ultrasound Med Biol. 2016 Feb;42(2):378-86. doi: 10.1016/j.ultrasmedbio.2015.10.003. Epub 2015 Nov 6. PMID 26553206
- [Background] Choi YJ, Lee JH, Lim HK, Kim SY, Han MW, Cho KJ, Baek JH. Quantitative shear wave elastography in the evaluation of metastatic cervical lymph nodes. Ultrasound Med Biol. 2013 Jun;39(6):935-40. doi: 10.1016/j.ultrasmedbio.2012.12.009. Epub 2013 Feb 27. PMID 23453381
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/